CLINICAL TRIAL: NCT05895604
Title: The Mother in Norway Study - A Randomised Trial of Nurse-Family Partnership (NFP)
Brief Title: The Mother in Norway Study
Acronym: MiNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other); Norwegian Institute of Public Health (Other Government); The Norwegian Directorate for Children, Youth and Family Affairs (Other); Norwegian Center for Violence and Traumatic Stress Studies (Other); Regional centre for children and youth mental health and welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NFP-202862
Record Dates: First submitted 2023-04-17; First posted 2023-06-08 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Maternal Behavior; Injuries; Violence; Mental Health Wellness
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment-NFP (Experimental): NFP is a prenatal and infancy home visiting program for vulnerable first-time mothers and their families. Registered nurses begin visiting their clients as early in the pregnancy as possible, guiding the mothers-to-be on different aspects of the parental role and offer practical and emotional support. The nurses continue visiting regularly until the child is two years old (up to 64 visits in total).
  Interventions: Behavioral: Nurse-Family Partnership
- Control (No Intervention): Control group members have access to the standard of care and whatever other programs and services are available in the community.

INTERVENTIONS:
Behavioral: Nurse-Family Partnership — Nurse-Family Partnership is a prenatal and infancy home visiting program providing regular visits to first-time mothers until the child is two years old
  Arms: Treatment-NFP

SUMMARY:
The Norwegian government is implementing the Nurse Family Partnership program (NFP) to combat child abuse and social inequality. This study will examine NFP with an individually randomized controlled parallel-group trial. The study will enroll 700 mothers over three years, with half receiving NFP services and the other half receiving standard care. The primary outcome is violence towards mothers and their children, assessed through questionnaires and observation tests. The study will also evaluate the program's effects on various health-related outcomes using administrative data. Cost-effectiveness analyses will be conducted to compare NFP to existing services and improve its delivery efficiency.

DETAILED DESCRIPTION:
The Norwegian government has since 2015 been in the process of implementing the Nurse Family Partnership program (NFP) in Norway, as a possibly important part in their strategy to combat child abuse and social inequality. This study employs an individually randomized controlled parallel-group trial where participants are randomly assigned to experimental and control groups. The planned study population consists of 700 mothers to be enrolled over 3 years (June 2023-2026). Each participant will be individually randomized with a 50 percent probability of being assigned to the treatment group, and a 50 percent probability of being assigned to the control group. NFP services will be provided to those in the treatment group through the child's second birthday (2025-2029). The control group will receive the standard of care and whatever other programs and services are available in the community.

Primary outcome is violence towards first-time mothers and their children. In their last trimester, and when the child is 6, 12 and 24 months old, mothers included in the study will receive a questionnaire assessing perceived partner violence, parenting skills, coping, control, and the child's development and language. At 24 months, staff at health stations will perform the Bayley observation test of the child´s development and language. The study will also utilise administrative data to assess the effects of NFP on a wide range of health- and health related outcomes. All analyses are carried out blinded. The investigators estimate "intention-to-treat" (ITT) effects and per-protocol analysis. Cost-effectiveness analyses will be conducted to compare the value of NFP to existing services, and to improve the efficiency in the delivery of NFP.

ELIGIBILITY:
Inclusion Criteria: Female; No previous live births; Currently pregnant; Gestation period less than 28 weeks (i.e., less than or equal to 27 weeks, 6 days) at time of recruitment; Live within an area serviced by a NFP Implementing Agency; Not currently enrolled in the study; professionals are concerned about the pregnancy / impending parenthood

Exclusion Criteria: Women who have had a previous live birth; Women who are not currently pregnant; Women who are past their 28th week of gestation (i.e., greater than or equal to 28 weeks, 0 days) at time of recruitment; Women who live outside of an area serviced by a NFP Implementing Agency; Women who are currently enrolled in the study; professionals are not concerned about the pregnancy / impending parenthood

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2042-12-31 (Estimated)

PRIMARY OUTCOMES:
Domestic violence (change is being assessed) | baseline, in last trimester, at 6, 12 and 24 months postpartum
  Composite Abuse Scale - Revised Short Form (CASr-SF). Items are scored on a scale ranging from 1-5, where higher scores indicate worse outcomes
Child maltreatment (change is being assessed) | at 12 and 24 months postpartum
  Brief Child Abuse Potential Inventory (BCAPI). Items are scored on a dichotomous range (agree/disagree), where higher scores indicate better outcomes
Child welfare service reports | 24 months postpartum
  Total number of reports to the child welfare service due to violence since birth
Child welfare service measures | 24 months postpartum
  Total number of provided measures and care takeovers due to violence since birth
Injuries (change is being assessed) | at delivery, 6, 12 and 24 months postpartum
  Hospital admissions

SECONDARY OUTCOMES:
Parental skills (change is being assessed) | at 6, 12 and 24 months postpartum
  Parenting Sense of Competence Scale (PSOC). Items are scored on a scale ranging from 1-6, where higher scores indicate better outcomes
Interaction between mother and child | at 12 months postpartum
  Emotional Availability Scale. Items are scored on a scale ranging from 1-7, where higher scores indicate better outcomes
Self-Efficacy (change is being assessed) | at baseline, and at 6, 12 and 24 months postpartum
  General Self-Efficacy Scale (GSE). Items are scored on a scale ranging from 1-4, where higher scores indicate better outcomes
Parental Locus of Control (change is being assessed) | at 6, 12 and 24 months postpartum
  Parental locus of control (PLOC). Items are scored on a scale ranging from 1-5, where lower scores indicating internal control and higher scores indicating external control
Child Development | at 24 months postpartum
  Bayley scale of infant development
Health-related Quality of Life (change is being assessed) | baseline, in last trimester, at 6, 12 and 24 months postpartum
  EQ-5D (the EuroQol Instrument), Items are scored on a scale ranging from 1-5, where higher scores indicate worse outcomes
Health behaviour (change is being assessed) | baseline, in last trimester, at 6, 12 and 24 months postpartum
  Use of tobacco, alcohol, drugs

CONTACTS AND LOCATIONS:
Overall Officials: Anne Grete Tøge, phd, Principal Investigator — Oslo Metropolitan University; Eirin Pedersen, phd, Principal Investigator — Oslo Metropolitan University
Locations (5):
- Norway (5):
  - Region Vestland, Bergen, Bergen
  - Region Agder, Kristiansand, Kristiansand
  - Region Rogaland, Sandnes, Sandnes
  - Region Trøndelag, Trondheim, Trondheim
  - Region Oslo, Oslo

IPD SHARING:
Plan to Share IPD: No